CLINICAL TRIAL: NCT00339144
Title: A Phase I Study of BMS-354825 in Patients With Solid Tumors
Brief Title: Study of Dasatinib (BMS-354825) in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-058
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Tumors
Keywords: Solid tumors (including relapsed disease) that are refractory to standard therapies or for which no effective standard therapy exists
MeSH Terms: conditions — Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dasatinib (100 mg) (Experimental)
  Interventions: Drug: Dasatinib
- Dasatinib (150 mg) (Experimental)
  Interventions: Drug: Dasatinib
- Dasatinib (200 mg) (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — tablets, Oral, 100 mg, once daily for 4 weeks
  Other Names: Sprycel; BMS-354825
  Arms: Dasatinib (100 mg)
Drug: Dasatinib — tablets, Oral, 150 mg, once daily, 4 weeks
  Other Names: Sprycel; BMS-354825
  Arms: Dasatinib (150 mg)
Drug: Dasatinib — tablets, Oral, 200 mg, once daily for 4 weeks
  Other Names: Sprycel; BMS-354825
  Arms: Dasatinib (200 mg)

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) or the maximum administered dose (MAD) of Dasatinib (BMS-354825) in patients in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Performance status (general conditions) specified by the Eastern Cooperative Oncology Group: 0-2
* Histologic or cytologic diagnosis of a solid tumor which has progressed on or following standard therapies (including relapsed disease) or for which no standard therapy exists.
* men and women, ages 20 and over
* women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 3 months after the study in such a manner that the risk of pregnancy is minimized
* Adequate hepatic function

Exclusion Criteria:

* Participants who are eligible and willing to undergo transplantation at pre- study.
* Women who are pregnant or breastfeeding with known brain metastasis or symptoms of brain metastasis
* Uncontrolled or significant bleeding disorder unrelated to a primary tumor
* Dementia or mental illness that would prohibit understanding or giving informed consent.
* Severe allergy to drugs required for appropriate supportive care of patients in this study.
* History of gastrointestinal surgery or of any digestive disorder which has the potential to inhibit absorption of the study drug.
* Pleural effusion > Grade 1
* Patient with dysphagia
* Does not agree to blood/blood products transfusion(s)
* Donated blood over 200 mL within 4 weeks prior to the start of study therapy
* Medication that known to have a risk of causing Torsade de pointes
* Participants who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Sayama, Osaka
  - Local Institution, Koto-Ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib 100 mg: Participants were administered an oral dose of 100 mg dasatinib tablet once daily for a period of 4 weeks. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level. Dose was not escalated above 200 mg daily.
- Dasatinib 150 mg: Participants were administered an oral dose of 150 mg dasatinib tablet once daily for a period of 4 weeks. Initially, 3 participants were treated at one dose level. If no DLT was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level. Dose was not escalated above 200 mg daily.
- Dasatinib 200 mg: Participants were administered an oral dose of 200 mg dasatinib tablet once daily for a period of 4 weeks. Initially, 3 participants were treated at one dose level. If no DLT was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. Dose was not escalated above 200 mg daily.
Period: Overall Study
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Started | 9 (Number of participants enrolled and treated) | 3 (Number of participants enrolled and treated) | 4 (Number of participants enrolled and treated)
Completed | 0 | 0 | 0
Not Completed | 9 | 3 | 4
Not completed — Disease progression | 5 | 2 | 2
Not completed — Study drug toxicity | 3 | 1 | 1
Not completed — Participant's request to discontinuation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg | Total
Number analyzed (Participants) | 9 | 3 | 4 | 16
Age Continuous [Median (Full Range); unit: years] | 58.0 [33.0 to 65.0] | 55.0 [39.0 to 63.0] | 47.5 [33.0 to 53.0] | 54.0 [33.0 to 65.0]
Age, Customized [Number; unit: participants]
  < 65 years | 7 | 3 | 4 | 14
  >=65 years | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 3 | 11
  Male | 2 | 2 | 1 | 5
Eastern Cooperative Oncology group (ECOG) Performance Status (PS) [Number; unit: Units on a scale] — The ECOG PS is used to assess disease severity. ECOG PS scores are, 0: fully active, able to carry on all pre-disease performance without restriction; 1: restricted physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3: capable of only limited self care, confined to bed or chair more than 50% of waking hours; 4: completely disabled, cannot carry on any self-care i.e. totally confined to bed or chair.
  Units on a scale
    0 = Fully active | 7 | 1 | 2 | 10
    1 = Ambulatory and able to work | 2 | 2 | 2 | 6
    2 = Ambulatory but unable to work | 0 | 0 | 0 | 0
    3 = Capable of only limited self care | 0 | 0 | 0 | 0
    4 = Completely disabled | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Maximum Acceptable Dose (MAD) of Dasatinib as Determined by Number of Participants With Dose-Limiting Toxicities (DLTs) Related to Dasatinib Treatment
Description: MAD: highest dose level at which >=1 DLTs were reported, MTD: dose one step lower than MAD. DLT: any of the following considered related to dasatinib during course 1:Grade 3(dose reduction by 1 dose level)/Grade 4:recurring nausea, vomiting or diarrhea; any other Grade >=3 non-hematologic toxicity except alopecia or fatigue;any grade toxicity requiring two dose reductions or participant's discontinuation; Grade 4 neutropenia <500 cells/mm^3 for >=5 consecutive days or febrile neutropenia; Grade 4 thrombocytopenia <25,000 cells/mm^3 or Grade 3 bleeding requiring platelet transfusion.
Time Frame: From start of the treatment i.e.Day 1 to end of Cycle 1 i.e. Day 30 (4 weeks)
Population: All treated participants who received at least one dose of the study drug and were evaluable for DLT.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 6 | 3 | 3
participants | 1 | 0 | 1

2. Secondary Outcome: Number of Participants Who Died, Experienced Adverse Events (AEs), Serious AEs (SAEs), Drug Related AEs and Discontinued Due to AEs
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to an AE were recorded. Drug-related AEs: events with a relationship to the study therapy of certain; probable; possible; not likely or unrelated.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All participants who received at least one dose of the study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants
  Deaths | 0 | 0 | 0
  AEs | 9 | 3 | 4
  SAEs | 1 | 1 | 1
  Drug-related AEs | 9 | 3 | 4
  All AEs Leading to Discontinuation | 3 | 1 | 1

3. Secondary Outcome: Number of Participants With Grade 3 or 4 Hematology Abnormalities
Description: Hematology abnormalities were graded per the National Cancer Institute (NCI) Common. Terminology Criteria (CTC) version 3.0 criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: Absolute Neutrophil Count (ANC): Grade 3: 0.5 - <1.0*10^9/L, Grade 4: <0.5*10^9/L; lymphocytes: Grade 3: 0.2 - <0.5*10^9/L, Grade 4: <0.2*10^9/L.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants
  Low neutrophils count | 1 | 0 | 0
  Low lymphocyte count | 0 | 1 | 2

4. Secondary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities
Description: Abnormalities were graded according to the NCI CTC, version 3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: phosphorous: Grade 3: 1.0-<2.0 mg/dL, Grade 4: <1.0 mg/dL; calcium: Grade 3: 6.0-<7.0 or >12.5-13.5 mg/dL, Grade 4: <0.6->13.5 mg/dL; magnesium: Grade 3: >3.0 - 8.0 mg/dL or >1.23 - 3.30 mmol/L, Grade 4: >8.0 mg/dL or >3.30 mmol/L; albumin: Grade 3: <2 g/dL or <20 g/L.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants
  Low phosphorus | 0 | 0 | 1
  Low calcium | 0 | 0 | 1
  High magnesium | 1 | 0 | 1
  Low albumin | 0 | 0 | 1

5. Secondary Outcome: Most Frequent Grade 3-4 Hematology Abnormalities Occurring in >=10% Participants: Low Lymphocyte Count
Description: Abnormalities were graded according to the NCI CTC, version 3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Most frequent hematology Grade 3 and 4 abnormalities occurring in >=10% participants were recorded. Grade 3 and 4 criteria are as follows: lymphocyte count: Grade 3: 0.2 - <0.5*10^9/L, Grade 4: <0.2*10^9/L.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants | 0 | 1 | 2

6. Secondary Outcome: Most Frequent Serum Chemistry Laboratory Abnormalities Occurring in >=10% Participants: High Magnesium
Description: Abnormalities were graded according to the NCI-CTC, version 3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Most frequent (>=10%) serum laboratory abnormalities were recorded. The following definitions specify the NCI-CTC AE criteria for serum laboratory abnormalities in the data presented: magnesium: Grade 3: >3.0 - 8.0 mg/dL or >1.23 - 3.30 mmol/L, Grade 4: >8.0 mg/dL or >3.30 mmol/L.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All participants who received at least one dose of the study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants | 1 | 0 | 1

7. Secondary Outcome: Number of Participants With Clinically Meaningful Physical Examination Measures
Description: Interim and final physical examinations were performed. The investigator used his/her clinical judgment to decide whether or not physical examination findings were clinically significant.
Time Frame: From screening, Day 1 in each treatment course and at the end of study
Population: All participants who received at least one dose of the study drug (safety population). Analysis for significant physical examination findings was not done.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Meaningful Vital Signs
Description: Vital signs measurements (including blood pressure, body temperature and pulse rate) were recorded. The investigator used his/her clinical judgment to decide whether or not abnormalities in vital signs were clinically significant.
Time Frame: From screening, Day 1 , 8, 15 and 22 in the 1st treatment course, Day 8 and 22 in the second and subsequent courses and at the end of study
Population: All participants who received at least one dose of the study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Standard 12-lead ECG was used to record selected ECG parameters like RR interval (the time between the two R waves in ECG), PR interval (interval measured from the beginning of the P wave to the beginning of the QRS complex; QRS complex is the name for some of the deflections seen on a typical ECG)), QRS duration, QT interval (time between onset of ventricular depolarization and end of ventricular repolarization), QT interval corrected for heart rate using Bazett's (QTcB) and Fridericia's (QTcF) formulas.
Time Frame: From screening Day -1, and at pre-dose, 1 and 4 hours (post-dose) on Days 1, 14 and 28 in first treatment course, at pre-dose, 1 and 4 hours (post-dose) during the second and fourth week in subsequent courses and at the end of study
Population: All participants who received at least one dose of the study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Change in QT Interval Corrected for Heart Rate (QTcF)
Description: QT interval corrected for heart rate (QTcF) was assessed using triplicate 12-lead serial ECGs.
Time Frame: Baseline, Day 1, Day 14 and Day 28
Population: All participants who received at least one dose of the study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants | 0 | 0 | 0

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Dasatinib
Description: Cmax was obtained from the plasma concentration versus time data after oral administration of dasatinib.
Time Frame: Blood samples were collected at 0 hour (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 12 and 24 hours (post dose) on Days 1, 14 and 28
Population: All treated participants with adequate pharmacokinetic (PK)profiles (PK population). The 'n' signifies those participants who received study drug and were evaluated for this measure (each group respectively).
Measure: Geometric Mean (Full Range); unit: nanograms (ng)/ml
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
nanograms (ng)/ml
  Day 1 (n = 9, 3, 4) | 139.83 [42.29 to 282.18] | 127.1 [73.30 to 308.42] | 124.48 [25.41 to 314.69]
  Day 14 (n = 5, 4, 2) | 137.03 [41.63 to 270.93] | 166.43 [59.21 to 651.67] | 102.61 [23.85 to 441.45]
  Day 28 (n= 3, 2, 2) | 253.77 [161.59 to 383.92] | 103.32 [35.40 to 301.52] | 80.92 [27.07 to 241.87]

12. Secondary Outcome: Area Under the Plasma-concentration-time Curve [AUC (INF)] of Dasatinib on Day 1
Description: AUC(INF), area under the plasma concentration-time curve from zero to the last time of the last quantifiable concentration within the dosing interval was calculated for Day 1.
Time Frame: Blood samples were collected at 0 hour (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 12 and 24 hours (post dose) on Day 1
Population: All treated participants with adequate PK profiles (PK population).
Measure: Geometric Mean (Full Range); unit: ng*hours/ml
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
ng*hours/ml | 537.98 [203.20 to 781.73] | 544.36 [346.36 to 962.79] | 595.62 [269.14 to 1166.52]

13. Secondary Outcome: AUC[TAU] of Dasatinib
Description: Area under the plasma concentration-time curve within the dosing interval was determined. AUC(TAU), from time 0 to the time of the last measurable concentration (24 hours) was calculated for Day 1, 14, 28 respectively.
Time Frame: as for outcome 11
Population: All treated participants with adequate PK profiles (PK population). The 'n' signifies those participants who received study drug and were evaluated for this measure (each group respectively).
Measure: Geometric Mean (Full Range); unit: ng*hours/ml
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
ng*hours/ml
  Day 1 (n = 9, 3, 4) | 524.55 [195.49 to 767.74] | 530.81 [338.10 to 953.62] | 528.65 [188.32 to 1123.34]
  Day 14 (n = 5, 4, 2) | 499.69 [217.19 to 681.86] | 694.90 [275.35 to 1798.79] | 716.27 [234.86 to 2184.52]
  Day 28 (n= 3, 2, 2) | 738.76 [497.44 to 1018.54] | 273.10 [150.69 to 494.93] | 534.33 [360.77 to 791.37]

14. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration of Dasatinib (Tmax)
Description: Tmax, time to reach maximum observed plasma concentration of dasatinib was obtained directly from the plasma concentration versus time data.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
hours
  Day 1 (n = 9, 3, 4) | 1.0 [0.5 to 4.0] | 1.0 [1.0 to 1.0] | 1.3 [0.5 to 3.0]
  Day 14 (n = 5, 4, 2) | 1.0 [0.5 to 3.0] | 1.0 [1.0 to 1.0] | 2.3 [1.5 to 3.0]
  Day 28 (n= 3, 2, 2) | 0.5 [0.5 to 1.0] | 0.5 [0.5 to 0.5] | 3.3 [0.5 to 6.0]

15. Secondary Outcome: Terminal Elimination Half-life (T-half) of Dasatinib
Description: T-half of dasatinib was calculated using plasma concentration versus time data.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
hours
  Day 1 (n = 9, 3, 4) | 4.77 (0.61) | 4.68 (0.84) | 7.62 (4.11)
  Day 14 (n = 5, 4, 2) | 5.75 (1.67) | 5.04 (0.19) | 7.95 (5.62)
  Day 28 (n= 3, 2, 2) | 4.36 (1.19) | 8.33 (2.78) | 7.66 (4.24)

16. Secondary Outcome: Accumulation Index (AI) of Dasatinib
Description: AI of Dasatinib was calculated as ratio of geometric mean of AUC(TAU) (area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration) on Day 14 or Day 28 on Day 1.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
ratio
  Day 14 (n = 5, 4, 2) | 0.81 [0.33 to 1.02] | 1.78 [1.42 to 2.11] | 2.30 [1.25 to 4.25]
  Day 28 (n= 3, 2, 2) | 1.12 [0.73 to 1.57] | 0.48 [0.45 to 0.52] | 1.72 [1.54 to 1.92]

17. Secondary Outcome: Mean Apparent Oral Clearance (CLo) of Dasatinib
Description: Apparent oral clearance was obtained from the plasma concentration versus time data.
Time Frame: Blood samples were collected at 0 hour (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 12 and 24 hours (post dose) on Days 14 and 28
Population: as for outcome 13
Measure: Geometric Mean (Full Range); unit: L/hour
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
L/hour
  Day 14 (n = 5, 4, 2) | 200.12 (134.3) [146.66 to 460.42] | 215.86 (204.7) [83.39 to 544.77] | 279.22 (537.4) [91.55 to 851.59]
  Day 28 (n= 3, 2, 2) | 135.36 (53.3) [98.18 to 201.03] | 549.26 (489.6) [303.07 to 995.41] | 374.30 (231.3) [252.73 to 554.37]

18. Secondary Outcome: Mean Apparent Volume of Distribution (Vz/F) of Dasatinib
Description: Apparent volume of distribution after oral dosing was obtained from plasma concentration versus time data.
Time Frame: as for outcome 17
Population: as for outcome 13
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
L
  Day 14 (n = 5, 4, 2) | 1156.57 (2010) [624.44 to 5283.67] | 1285.05 (1967) [437.91 to 4780.03] | 2903.18 (12216) [474.80 to 17751.50]
  Day 28 (n= 3, 2, 2) | 566.93 (286) [425.51 to 935.66] | 3443.56 (5920) [1234.38 to 9606.51] | 3362.08 (6081) [1158.35 to 9758.36]

19. Secondary Outcome: Cmax of Metabolite BMS-582691
Description: Maximum plasma concentration was obtained from plasma concentration versus time data of metabolite (BMS-582691).
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Full Range); unit: ng/ml
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
ng/ml
  Day 1 (n = 8, 3, 3) | 5.18 [1.93 to 11.93] | 2.89 [1.11 to 8.33] | 7.90 [4.83 to 11.91]
  Day 14 (n = 5, 4, 2) | 4.63 [1.26 to 11.13] | 4.61 [2.29 to 14.94] | 5.99 [1.51 to 23.74]
  Day 28 (n= 3, 1, 2) | 6.68 [4.26 to 9.35] | 4.66 [4.66 to 4.66] | 3.04 [1.17 to 7.91]

20. Secondary Outcome: AUC (0-t) of Metabolite BMS-582691
Description: AUC (0-t) was calculated using plasma concentration values of metabolite at time 0 to the time of the last measurable concentration (t).
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
ng*hr/mL
  Day 1 (n = 8, 3, 3) | 21.24 [12.10 to 40.55] | 5.99 [0.55 to 29.00] | 36.96 [28.68 to 50.78]
  Day 14 (n = 5, 4, 2) | 15.24 [2.02 to 35.05] | 26.05 [8.92 to 84.33] | 37.65 [9.35 to 151.70]
  Day 28 (n= 3, 1, 2) | 27.20 [22.85 to 35.47] | 13.03 [13.03 to 13.03] | 4.67 [0.59 to 37.23]

21. Secondary Outcome: Tmax of the Metabolite BMS-582691
Description: Tmax of the metabolite was obtained using plasma concentration versus time data of metabolite BMS-582691.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
hours
  Day 1 (n = 8, 3, 3) | 1.5 [1.0 to 4.0] | 1.5 [1.0 to 1.5] | 2.0 [1.5 to 2.0]
  Day 14 (n = 5, 4, 2) | 1.0 [1.0 to 3.0] | 1.8 [1.5 to 3.0] | 3.0 [3.0 to 3.0]
  Day 28 (n= 3, 1, 2) | 1.5 [1.0 to 1.5] | 1.0 [1.0 to 1.0] | 1.8 [1.5 to 2.0]

22. Secondary Outcome: Mean Urine Concentration of Urinary N-telopeptide Type 1 Collagen (NTx) Biological Marker
Description: Urine NTx is a measure of bone metabolism. A decrease in the marker relative to baseline indicates a decrease in bone metabolism. Mean urine concentration of NTx biological marker was determined using enzyme linked immuno-sorbent assay (ELISA).
Time Frame: Urine samples were collected at baseline (Day -1) and 0 hour (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 12 and 24 hours (post dose) on Days 14 and 28.
Population: All treated participants with adequate pharmacodynamic (PD) profiles (PD population). The 'n' signifies those participants who received study drug and were evaluated for this measure (each group respectively).
Measure: Mean (Standard Deviation); unit: nmol*bone collagen equivalent (BCE)/mmol
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
nmol*bone collagen equivalent (BCE)/mmol
  Day -1 ( n= 9, 3, 4) | 51.71 (39.75) | 62.57 (15.78) | 103.90 (57.37)
  Day 14 (n= 6, 3, 4) | 51.55 (59.74) | 36.47 (26.00) | 51.33 (30.08)
  Day 28 (n= 3, 2, 2) | 25.33 (4.26) | 40.10 (16.40) | 36.15 (36.84)

23. Secondary Outcome: Mean Urine Concentration of Deoxypyridinoline (Dpyr) Biological Marker
Description: Urine levels of DPyr is a measure of bone resorption. A decrease in Dpyr relative to the baseline indicates decrease in bone metabolism. Mean urine concentration of Dpyr biological marker was determined using ELISA.
Time Frame: Urine samples were collected at baseline (Day -1) and 0 hour (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6 12 and 24 hours post dose on Days 14 and 28
Population: All treated participants with adequate PD profiles (PD population). The 'n' signifies those participants who received study drug and were evaluated for this measure (each group respectively).
Measure: Mean (Standard Deviation); unit: nanomol (nmol)/mL
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
nanomol (nmol)/mL
  Day -1 (n = 9, 3, 4) | 37.79 (50.04) | 50.37 (54.05) | 116.85 (134.73)
  Day 14 (n= 6, 3, 4) | 27.08 (32.15) | 25.37 (25.22) | 46.73 (47.24)
  Day 28 (n= 3, 2, 2) | 15.77 (17.34) | 40.55 (37.97) | 14.80 (14.14)

24. Secondary Outcome: Mean Serum Concentration of Tartrate-resistant Acid Phosphatase Isoform 5b (TRACP-5b) Biological Marker
Description: TRACP-5b is a measure of bone metabolism. A decrease in TRACP-5b relative to the baseline indicates decrease in bone metabolism. Serum TRACP-5b was quantified with enzyme-linked-immunosorbent serologic assay (ELISA).
Time Frame: Serum samples were assessed at baseline (Day -1) and on Days 14 and 28
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Dasatinib (Total): Dasatinib(100 mg, 150 mg, 200 mg) was administered once daily via oral route for a period of 4 weeks. Initially, 3 participants were treated at one dose level. If no DLT was observed, the dose would be escalated to next higher level. If a DLT was observed among one of three treated participants in the first course at a dose level, 3 participants would be additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose might be escalated to next higher dose level.
Arm/Group | Dasatinib (Total)
Number analyzed (Participants) | 16
U/L
  Day -1 (n = 16) | 5.13 (1.89)
  Day 14 (n= 12) | 4.13 (1.25)
  Day 28 (n= 7) | 3.40 (0.61)

25. Secondary Outcome: Mean Serum Concentration of Bone Alkaline Phosphatase (BAP) Biological Marker
Description: BAP is a measure of bone metabolism. A decrease in BAP relative to the baseline indicates decrease in bone metabolism. Serum BAP was quantified with ELISA.
Time Frame: Serum samples were assessed on baseline (Day -1), and pre-dose on Days 14, 28
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dasatinib (Total)
Number analyzed (Participants) | 16
U/L
  Day -1 (n = 16) | 29.11 (11.21)
  Day 14 (n= 13) | 32.34 (11.92)
  Day 28 (n= 7) | 28.20 (6.21)

26. Secondary Outcome: Number of Participants With Sarcoma (Src) and Phosphorylated Src (pSRc) Protein Expression in Peripheral Blood Mononuclear Cells (PBMC)
Description: Src and pSrc protein expression was planned to be evaluated in PBMC for establishing PK/PD relationship between Src/pSrc protein expression in PBMC and exposure of BMS-354825.
Time Frame: Plasma samples were collected on baseline (Day -1), 0 hour (pre-dose), 1 and 4 hours (post-dose) on Days 1, 14 and 28
Population: All treated participants with adequate pharmacodynamic profiles. Participants could not be evaluated as the test was discontinued due to difficulty in appropriate measurements.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: Tumor response was defined as the number of participants whose best response was CR or PR as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR: disappearance of all target/non-target lesions; PR: >= 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Within 4 weeks of first study drug administration, thereafter recorded every 4 or 8 weeks.
Population: All treated participants with measurable disease at baseline and received at least one dose of the study drug (efficacy population).
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Number analyzed (Participants) | 9 | 3 | 4
participants
  CR | 0 | 0 | 0
  PR | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dasatinib 100 mg | Dasatinib 150 mg | Dasatinib 200 mg
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/3 | 1/4
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg (N=9) | Dasatinib 150 mg (N=3) | Dasatinib 200 mg (N=4)
Perianal abscess (Infections and infestations) | 1 | 0 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg (N=9) | Dasatinib 150 mg (N=3) | Dasatinib 200 mg (N=4)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 4
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Conjunctival hemorrhage (Eye disorders) | 1 | 0 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 2 | 2
Nausea (Gastrointestinal disorders) | 5 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Painful defecation (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 2 | 4
Edema (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Face edema (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Peripheral coldness (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1
Blood calcium decreased (Investigations) | 2 | 1 | 2
White blood cell count decreased (Investigations) | 4 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1
Blood urine present (Investigations) | 2 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 2
Protein urine (Investigations) | 1 | 0 | 2
Blood phosphorus decreased (Investigations) | 0 | 1 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0
Blood magnesium increased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 2 | 0 | 0
Blood sodium decreased (Investigations) | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1
Hemoglobin decreased (Investigations) | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 2
Red blood cell count decreased (Investigations) | 2 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Hematocrit decreased (Investigations) | 1 | 0 | 0
Prothrombin time ratio increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1
Cell marker increased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Breast hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Nipple swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.